CLINICAL TRIAL: NCT01574508
Title: Continuous Subcutaneous Insulin Infusion strAtegy Versus Multiple Daily Insulin Injections strAtegy
Acronym: CAMACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD012
Record Dates: First submitted 2012-01-25; First posted 2012-04-10 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Type 2 Diabetes
Keywords: efficacy; safety; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Continuous Subcutaneous Insulin Infusion (Experimental): CSII
  Interventions: Drug: Transient Continuous Subcutaneous Insulin Infusion
- Multiple Daily Insulin Injections (Active Comparator): MDI
  Interventions: Drug: Transient Multiple Daily Insulin Injections

INTERVENTIONS:
Drug: Transient Continuous Subcutaneous Insulin Infusion — Patients will be given Continuous Subcutaneous Insulin Infusion during two weeks confinement in the hospital. The initial dosage will be body weight (kg)*0.5, and will be adjusted according to the 7 points glucose monitoring records in the hospital.
  Other Names: CSII
  Arms: Continuous Subcutaneous Insulin Infusion
Drug: Transient Multiple Daily Insulin Injections — Patients will be given Transient multiple daily insulin injections during two weeks confinement in the hospital. The initial dosage will be body weight (kg)*0.5, and will be adjusted according to the 7 points glucose monitoring records in the hospital
  Other Names: MDI
  Arms: Multiple Daily Insulin Injections

SUMMARY:
The current study will compare the different efficacy of two transient intensive insulin treatment strategies: Continuous subcutaneous insulin infusion (CSII) and multiple daily insulin injections (MDI) in patients who are not well controlled with oral hypoglycaemic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Using at least two kinds of oral hypoglycaemic agents, one of which must be insulin secretagogues (at least half of the maximum permitted daily dose); or at least two kinds of oral hypoglycaemic agents, one of which must be insulin secretagogues (at least half of the maximum permitted daily dose), plus once daily basic insulin treatment (daily dosage < 30IU);
2. The anti-diabetic therapy is stable within 3 months before study screening;
3. Age: 25-65years, both gender, BMI: 20-35kg/m2;
4. Good compliance with the follow-up
5. Signed informed consent
6. HbA1c ≥ 8.0 % and ≤ 12%

Exclusion Criteria:

1. Having the history of using insulin therapy twice daily or MDI or insulin pump (except the insulin therapy during gestational diabetes mellitus)
2. For once daily insulin therapy: daily dose insulin therapy dosage > 30IU
3. Having the history of using GLP-1 for therapy within 3 months before screening
4. Women in pregnancy or under breast feeding
5. Having acute diabetic complications within 6 months before screening or having severe chronic diabetic complications at screening
6. Allergic to study drugs
7. Severe liver dysfunction, including serum alanine aminotransferase concentration more than 2.5 times above upper limit of normal range, abnormal renal function (GFR < 60ml/min)
8. Other severe conditions which will put the patients in high risk during the study
9. Recently drug or alcohol abuse

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin levels | During 2 weeks intensive insulin treatment period and 1 year after the intensive treatment.
  The different influence of two intensive insulin treatment strategies: CSII and MDI on the change of glycated hemoglobin levels during two weeks intensive insulin treatment period and 1 year after the intensive treatment.
Glycated albumin levels | During 2 weeks intensive insulin treatment period and 1 year after the intensive treatment.
  The different influence of two intensive insulin treatment strategies: CSII and MDI on the change of glycated albumin levels during two weeks intensive insulin treatment period and 1 year after the intensive treatment.

SECONDARY OUTCOMES:
The glucose levels | During 2 weeks intensive treatment and 1 year after treatment
  The different influence of CSII and MDI on the change of plasma glucose levels during 2 weeks intensive treatment and 1 year after treatment
Episode of hypoglycemia | During 2 weeks of intensive treatment and 1 year after treatment
  The different influence of CSII and MDI on Episode of hypoglycemia during 2 weeks of intensive treatment and 1 year after treatment
Body weight | During 2 weeks intensive treatment and 1 year after treatment
  The different influence of CSII and MDI on Body weight during 2 weeks intensive treatment and 1 year after treatment
Biochemical parameters and inflammatory factors | During 2 weeks intensive treatment and 1 year after treatment
  The different influence of CSII and MDI on the change of biochemical parameters and inflammatory factors during 2 weeks intensive treatment and 1 year after treatment
C peptide levels | During 2 weeks intensive treatment and 1 year after treatment
  The different influence of CSII and MDI on the change of C peptide levels during 2 weeks intensive treatment period and 1 year after treatment
Number of participants with adverse events | During 2 weeks intensive treatment and 1 year after treatment
  The number of Participants with adverse events in different intensive treatment strategies (CSII or MDI) during 2 weeks intensive treatment period and 1 year after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China